CLINICAL TRIAL: NCT02174068
Title: A Pharmacokinetic Drug Interaction and Tolerance Study of Paracetamol and Nefopam
Acronym: PARA-NEF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0191; 2014-000624-22
Record Dates: First submitted 2014-05-26; First posted 2014-06-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
Keywords: Paracetamol; Nefopam; Pharmacokinetic; Drug interaction
MeSH Terms: interventions — Acetaminophen; Nefopam

ARMS (1):
- paracetamol (Experimental): drug interaction between paracetamol and nefopam in healthy volunteers.
  Interventions: Drug: paracetamol 1000 mg per os, nefopam 60mg per os, paracetamol 1000 mg + nefopam 60 mg per os

INTERVENTIONS:
Drug: paracetamol 1000 mg per os, nefopam 60mg per os, paracetamol 1000 mg + nefopam 60 mg per os

SUMMARY:
Pain remains the leading cause of consultation. Despite a wide therapeutic arsenal, a significant percentage of patients disclaim little or no pain relief with common analgesics, specific or not their type of pain. This is especially true in cases of chronic pain, and current treatments are associated with many side effects. A need for therapeutic innovation is needed. Paracetamol is currently the most widely used analgesic worldwide but despite its excellent safety, its analgesic effect is limited from moderate to severe pain. Many analgesic drug combinations include paracetamol, recently the co-administration of paracetamol and nefopam showed a supra-additive antinociceptive effect (Van Elstraete AC et al. 2013). The development of a formulation associating paracetamol and nefopam first requires searching a possible pharmacokinetic interaction between the two active substances and assessing safety of this combination in healthy volunteers. No published studies providing such information.

DETAILED DESCRIPTION:
This is a randomised, cross-over, open label trial assessing drug interaction between paracetamol and nefopam in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* ALT, AST, PAL, normal GGT, creatinine <133μmol / L, hematocrit>38%
* Informed consent to the trial
* Healthy volunteers affiliated to the French Social Security

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Existence of drug interaction | AT DAY 1
  Drug metabolites and principle assessing by LC / MS / MS in blood samples. Determining of Cmax, Tmax, AUC and Half-life

SECONDARY OUTCOMES:
influence of paracetamol on the kinetics of nefopam | AT DAY 1
Measure of plasma pharmacokinetic parameters of each active metabolites and principles (dosage nefopam, N-desmethyl-nefopam, paracetamol, paracetamol glucuronide, paracetamol sulfate) alone | at day 1
Measure of plasma pharmacokinetic parameters in combination (AUC, Cmax, Tmax, half-life time of apparent elimination terminal). | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France